CLINICAL TRIAL: NCT01929733
Title: Long Term Results of 450 Percutaneous Closures of PDA in a Single Center
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0192-13
Record Dates: First submitted 2013-08-14; First posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous closure is one of the methods used to treat, among other congenital heart disorder, Persistent Ductus Arteriosus (PDA) in children and adults. During the years 1998-2013 four hundred and fifty patients were catheterized in the department of pediatric cardiology and congenital heart diseases in Rambam health care campus, using various devices.

In this retrospective research, the investigators analyze data from patients' medical files, to estimate and define the correlation between the patients' demographic and morphologic data to the type and size of chosen closure device.

Aim of study:

To create an algorithm that can be used to choose the proper device for percutaneous closure of the PDA, based on the characteristics of the patient and the PDA type.

DETAILED DESCRIPTION:
The investigators analyze the demographic characteristics of patients before the procedure (Age, gender, weight, height, co-morbidities etc.), the type and characteristics of PDA and the chosen device, success and failure rates of the procedure, and adverse effects.

The data is taken from patients' medical files - based on medical reports regarding physical examination, blood tests and imaging studies including cineangiograms and echo-doppler studies.

ELIGIBILITY:
Inclusion Criteria:

* All the patients that underwent percutaneous closure of PDA between January 1998 and august 2013 in the department of pediatric cardiology and congenital heart diseases in Rambam health care campus

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients that underwent percutaneous closure of PDA between January 1998 and august 2013 in the department of pediatric cardiology and congenital heart diseases in Rambam health care campus
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 1998-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Success of implantation | one day, 10 days and a year after PDA closure and then last check-up exam
  due to the fact that the research is retrospective and refers to a period of 15 years (1998-2013)and the fact that some patients had a check-up exam from time to time - the investigators have decided to include in this research the last check-up exam as well.

SECONDARY OUTCOMES:
residual shunt | one day, 10 days and a year after PDA closure and then last check-up exam
  due to the fact that the research is retrospective and refers to a period of 15 years (1998-2013) and the fact that some patients had a check-up exam from time to time - the investigators have decided to include in this research the last check-up exam as well.

OTHER OUTCOMES:
Early and late Adverse effects | one day, 10 days and a year after PDA closure and then last check-up exam
  hemolysis, bleeding, infections ect. due to the fact that the research is retrospective and refers to a period of 15 years (1998-2013)and the fact that some patients had a check-up exam from time to time - the investigators have decided to include in this research the last check-up exam as well.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Dotan, MD, Principal Investigator — Rambam Health Care Campus; Omer Ephrat, Principal Investigator — Rambam Health Care Campus
Locations (1):
- RAMBAM health care center, Haifa, Israel